CLINICAL TRIAL: NCT01408082
Title: A Randomized, Double-Masked, Parallel-Group, Comparative Study to Evaluate the Clinical Efficacy and Safety of ISV-502 Compared to AzaSite Alone, Dexamethasone Alone, and Vehicle in the Treatment of Subjects With Non-Bacterial Blepharitis
Brief Title: Efficacy and Safety Study of a Steroid/Antibiotic Combination Eyedrop to Treat Non-Bacterial Blepharitis
Acronym: DOUBle
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-10-502-004
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis | interventions — Azithromycin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- ISV-502 (Experimental)
  Interventions: Drug: ISV-502 (1.0% azithromycin and 0.1% dexamethasone combined)
- AzaSite (Active Comparator)
  Interventions: Drug: Azasite
- Dexamethasone (Active Comparator)
  Interventions: Drug: Dexamethasone
- Vehicle (Placebo Comparator)
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: ISV-502 (1.0% azithromycin and 0.1% dexamethasone combined) — Azithromycin and Dexamethasone twice daily for 2 weeks
  Other Names: AzaSite Plus
  Arms: ISV-502
Drug: Azasite — Azasite twice daily for 2 weeks
  Arms: AzaSite
Drug: Dexamethasone — Dexamethasone twice daily for 2 weeks
  Arms: Dexamethasone
Other: Vehicle — Vehicle twice daily for 2 weeks
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of ISV-502 compared to AzaSite® alone, Dexamethasone alone, and vehicle in the treatment of subjects with Non-bacterial Blepharitis.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age at Visit 1 (Day 1, Baseline) of either sex and any race.
* Signature of the subject or legally authorized representative on the Informed Consent Form.
* Are willing and able to follow all instructions and attend all study visits.
* Are willing to avoid disallowed medication for the duration of the study.
* If female is of childbearing potential, agree to and submit a urine sample for pregnancy testing. Post menopausal is defined as having no menses for at least 12 consecutive months.
* Additional inclusion criteria also apply.

Exclusion Criteria:

* Have known sensitivity or poor tolerance to any component of the Investigational Drug.
* Have an acute ocular infection (bacterial, viral or fungal) or active ocular inflammation other than Blepharitis in the study eye.
* Have used topical corticosteroid medications or topical ophthalmic solutions that the investigator feels may interfere with the study parameters.
* Have used any non-diagnostic topical ophthalmic solutions in the study eye.
* Be currently pregnant, nursing, or planning a pregnancy; or be a woman that has a positive urine pregnancy test.
* Currently suffer from alcohol and/or drug abuse.
* Have prior (within 30 days of beginning dosing) or anticipated concurrent use of an investigational drug or device.
* Have a condition or a situation which, in the Investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation.
* Additional exclusion criteria also apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 917 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Clinical Resolution | Day 15
  The primary efficacy endpoint for the comparison of ISV-502 and AzaSite is complete clinical resolution of signs and symptoms at Day 15.
Recurrence of Clinical Signs and Symptoms | 6 Month
  The primary efficacy endpoint for the comparison of ISV-502 and Dexamethasone is recurrence of clinical signs and symptoms by 6-Month Follow-up.

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - Arizona Eye Center, Chandler, Arizona
  - Arizona Center for Clinical Trials LLC, Phoenix, Arizona
  - Cornea Consultants of Arizona, Phoenix, Arizona
  - Lugene Eye Institute, Glendale, California
  - United Medical Research Institute, Inglewood, California
  - Macy Eye Center, Los Angeles, California
  - North Valley Eye Medical Group, Inc., Mission Hills, California
  - Eye Research Foundation, Newport Beach, California
  - North Bay Associates, Inc., Petaluma, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Shasta Eye Medical Group, Inc., Redding, California
  - San Diego Eye and Laser Center, San Diego, California
  - West Coast Eye Care Associates, San Diego, California
  - Florida Eye Microsurgicial Institute, Inc., Boynton Beach, Florida
  - ZASA Clinical Research, LLC, Boynton Beach, Florida
  - Magruder Eye Institute, Orlando, Florida
  - Vision Eye Care Center, Palm Springs, Florida
  - International Research Center, Tampa, Florida
  - Richard Eiferman, MD, Louisville, Kentucky
  - Lakeview Optical, Gretna, Louisiana
  - Center for Sight, Inc., Fall River, Massachusetts
  - Tauber Eye Center, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Comprehensive Eye Care Ltd, Washington, Missouri
  - Abrams Eye Institute, Las Vegas, Nevada
  - Nevada Eye Care Professionals, Las Vegas, Nevada
  - Eye Care Associates of Nevada, Sparks, Nevada
  - David Ringel, OD PA, Sewell, New Jersey
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - Ophthalmic Consultants of Long Island, Valley Stream, New York
  - South Shore Eye Care, Wantagh, New York
  - Charlotte Eye Ear Nose & Throat Associates, P.A., Charlotte, North Carolina
  - Mundorf Eye Center, Charlotte, North Carolina
  - James Branch, MD, Winston-Salem, North Carolina
  - Eye Care Associates of Greater Cincinnati, Inc., Cincinnati, Ohio
  - Eye Care Associates of Greater Cincinnati, Inc., Fairfield, Ohio
  - Eye Care Associates of Greater Cincinnati, Inc., Madeira, Ohio
  - Roseburg Research Associates, LLC, Roseburg, Oregon
  - Philadelphia Eye Associates, Philadelphia, Pennsylvania
  - Research Across America @ Wyomissing Optometric Center Inc, Wyomissing, Pennsylvania
  - Total Eye Care, PA, Memphis, Tennessee
  - David Shulman, MD, San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - Daynes Eye and Lasik, Salt Lake City, Utah

REFERENCES:
- [Derived] Hosseini K, Bourque LB, Hays RD. Development and evaluation of a measure of patient-reported symptoms of Blepharitis. Health Qual Life Outcomes. 2018 Jan 11;16(1):11. doi: 10.1186/s12955-018-0839-5. PMID 29325546